CLINICAL TRIAL: NCT06735742
Title: TALZENNA Capsules Special Investigation - Investigation on BRCA Mutation-Positive and HER2-Negative Unresectable or Recurrent Breast Cancer With a History of Cancer Chemotherapy -
Brief Title: A Study to Learn About the Safety of TALZENNA for the Treatment of Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3441045
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: BRCA mutation-positive and HER2-negative; unresectable or recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to learn about the safety of TALZENNA for the patients with breast cancer that cannot be removed by surgery and has come back. These participants also have a past treatment with medicines that try to stop the growth of cancer cells.

This study is seeking for participants who:

* have breast cancer that cannot be removed by surgery and has come back
* have not used this medicine before. All patients in this study will receive TALZENNA according to the prescriptions.

Patients will be followed up to 52 weeks (12 months) from the day of start of treatment start (Day 1). However, in cases where treatment has been completed or stopped less than 52 weeks (12 months) after the start of giving study medicine, the participants will be checked until completion (discontinuation) of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BRCA mutation-positive and HER2- negative unresectable or recurrent breast cancer with a history of cancer chemotherapy
* No history of previous use of this drug

Exclusion Criteria:

* None

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who satisfy the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2025-04-12 (Actual); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions | Up to 52 weeks
  For adverse drug reactions corresponding to myelosuppression, interstitial lung disease, thromboembolism, and secondary malignant tumour, the incidence, time of onset, grade, outcome etc. will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Japan, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3441045